CLINICAL TRIAL: NCT01292408
Title: Autophagy Inhibition Using Hydrochloroquine in Breast Cancer Patients:a Pilot Study
Brief Title: Autophagy Inhibition Using Hydrochloroquine in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO201004
Record Dates: First submitted 2010-12-15; First posted 2011-02-09 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: autophagy; hydroxychloroquine; hypoxia; proven invasive adenocarcinoma of the breast: tumors are found to be ER negative (<10% ER pos cells)
MeSH Terms: conditions — Breast Neoplasms; Hypoxia | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily HCQ (Experimental): Between tumor biopsy and surgery, during 2-3 weeks, breast cancer patients will take daily HCQ, an anti-malaria and anti-rheumatic drug that precludes tumor cells from surviving hypoxia by inhibiting the process of autophagy in these cells
  Interventions: Drug: Hydrochloroquine

INTERVENTIONS:
Drug: Hydrochloroquine — 800 mg per os once, and then 400 mg per day
  Other Names: Plaquenil

SUMMARY:
Hydroxychloroquine is a drug that has been used to treat malaria and rheumatism. It is recently discovered that Hydroxychloroquine increases 'autophagy'. Autophagy is a process whereby cells eat a part themselves giving them extra energy. Cancer cells use autophagy to survive chemotherapy or hormonal therapy. Also, cancer cells use autophagy to survive in areas of a tumor where there is a low oxygen level.

The purpose of this study is to determine whether treatment with the drug Hydroxychloroquine leads to a decrease of autophagy in breast cancer tissue.

DETAILED DESCRIPTION:
In response to various stresses, cells can launch a process of "self-eating", termed autophagy. Thereby, components of the cell are catabolically digested via specific lysosomes called autophagosomes, to provide the cell with energy and other necessary factors to serve as a temporary survival mechanism (Chen et al. 2010).

Two major stressors that can be evaded by autophagy are important for cancer progression and treatment sensitivity:

1. cells can respond with autophagy to cytotoxic treatment such as chemo- or endocrine therapy, thereby leading to treatment insensitivity (Kondo et al. 2005; Chen et al. 2010), and
2. cells can survive severe hypoxia using autophagy (Rouschop et al. 2010), and hypoxic cells themselves are refractory to chemo-, endocrine and radiotherapy.

Thus, tumor cells evade treatment induced cell death by launching a temporary last survival mechanism. Inhibition of this pathway could lead to sensitization for a variety of cancer treatment regimen, or to specific cell killing of tumor associated hypoxic cells that would otherwise be refractory to radiotherapy. Chloroquine (CQ), N'-(7-chloroquinoline-4-yl)-N,N-diethyl-pentane-1,4-diamine, was discovered in 1934, and has widely been used as an effective and safe anti-malarial and anti-rheumatoid agent since 1947. Later, CQ has been rediscovered as a sensitizer of cytotoxic cancer therapies such as ionizing radiation and chemotherapeutics, although the precise mechanism behind this has remained largely unknown (Solomon and Lee 2009). Most recently, it was discovered that CQ inhibits the process of autophagy by impairment of autophagic vesicle clearance, as CQ accumulates in lysosomal vesicles. This has now lead to several investigators proposing that CQ or one of its analogs can be used to inhibit the autophagic pathway as an additive to other cytotoxic treatments. Hydrochloroquine (HCQ, Plaquenil) is a CQ derivative with fewer side effects than CQ, which has long been used as anti-malarial and antirheumatoid agent. It can be safely used at high doses for extended periods of time. Both CQ and HCQ are under investigation in clinical trials for glioblastoma, small and non-small cell lung cancer, breast cancer, prostate cancer, melanoma, renal cell carcinoma, and pancreatic cancer (for reviews see Solomon and Lee 2009 and Chen et al. 2010).

However, the effect of HCQ on tumor tissue, autophagy and/or oxygenation has of yet not been studied in human patients in vivo.

In this pilot study we intend to investigate the effect of HCQ on breast cancer tissues. To this end, breast cancer patients that have given informed consent for participation in the AFTER study (AMO 2010/312), but are not included as their tissue biopsy is found to be ER/PgR negative, will be asked to take 800 mg once, and then 400 mg/day HCQ for 2 to 3 weeks until surgery. We will compare tissue characteristics before and after treatment using HCQ, looking at effects on markers for both hypoxia and autophagy using immunohistochemistry. We expect that after treatment with HCQ tumor cells in hypoxic areas will no longer be able to survive, thus decreasing the number of viable hypoxic cells and increasing the amount of necrosis. This pilot study will serve as a proof of principle for future studies into the effect of autophagy inhibition on treatment sensitivity in breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with core-biopsy proven invasive adenocarcinoma of the breast
* Any tumor with a size ≥ 1cm (NOT inflammatory breast cancer)
* WHO-performance score 0 or 1
* Written informed consent

Exclusion Criteria:

* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol
* Hampered liver or kidney function
* Serious gastro-intestinal disease
* Neurological disease (including epilepsy)
* Hematological disease
* Psoriasis
* Porphyry
* G6PD deficiency
* Hypersensitivity for quinine
* Use of gold containing drugs, oxyphenbutazone, phenylbutazon, digoxin
* Operation for breast cancer foreseen within 14 days after inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
hypoxia markers | before and after short-term pre-surgical treatment with HCQ
  differences in endogenous hypoxia markers (CA9, PAI-1, VEGF [Rademakers et al. 2008]) and autophagy (LC3b [Rouschop et al. 2010]) before and after treatment with HCQ. These parameters will be quantified by immunohistochemistry on formalin fixed paraffin embedded tissue from both pretreatment biopsy, and posttreatment surgically obtained material.

SECONDARY OUTCOMES:
autophagy pathway mediators | before and after short-term pre-surgical treatment with HCQ
  differences in putative crucial mediators in the autophagy pathway currently under investigation, i.e. TRB3, ATF4, GRP78, LAMP3, etc.before and after short-term pre-surgical treatment with HCQ

CONTACTS AND LOCATIONS:
Overall Officials: P. Span, Md, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands